CLINICAL TRIAL: NCT06956560
Title: Microdosing, Non-randomized, Clinical Trial to Investigate Binding of Positron Emission Tomography Tracer [68ga]Ga-DOTA-Cys-ATH001 Targeting Platelet-derived Growth Factor Receptor Beta (PDGFRß) in Healthy Subject as Compared to Patients With Cardiac Fibrosis.
Brief Title: Platelet Derived Growth Factor Receptor ß (PDGFRß) Imaging in Cardiac Fibrosis
Acronym: PARIS
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: PARIS
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: ST-Elevation Myocardial Infarction (STEMI); Heart Failure With Preserved Ejection Fraction (HFpEF)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples for the future determination of exploratory biomarkers prior to administration of the PET-tracer will be collected at screening and at each PET examination.
  Biomarkers to be analyzed will include, but are not limited to: Nt-proBNP, Collagen I and III, C-terminal propeptide of procollagen type I (PICP), procollagen type I N-terminal propeptide (PINP), ProC3, procollagen type III amino-terminal propeptide (PIIINP), matrix metalloproteinases (MMPs)(e.g. MMP-1, MMP-2, MMP7…), tissue inhibitors of metalloproteinase (TIMPs) (e.g. TIMP1, TIMP-4…), transforming growth factor-β (TGF-β), connective tissue growth factor (CTGF), galectin-3 (Gal-3), pro-inflammatory mediators (tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β), IL-4, and IL-6…), microRNA (miR-1, miR-21…).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Individuals with high risk of heart failure after STEMI: Individuals with high risk of heart failure after STEMI are examined by PET using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan) at one week after PCI/stent intervention and at 2-8 months after PCI/stent.
  Interventions: Radiation: PET/MRI or separate PET/CT and MRI
- Individuals with low risk of heart failure after STEMI: Individuals with low risk of heart failure after STEMI are examined by PET using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan) at one week after PCI/stent intervention and at 2-8 months after PCI/stent.
  Interventions: Radiation: PET/MRI or separate PET/CT and MRI
- Individuals diagnosed with HFpEF and with signs/symptoms of heart failure: Individuals diagnosed with HFpEF are examined by PET using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan) once after inclusion.
  Interventions: Radiation: PET/MRI or separate PET/CT and MRI
- Healthy control individuals: Healthy control individuals are examined by PET using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan) once after inclusion.
  Interventions: Radiation: PET/MRI or separate PET/CT and MRI

INTERVENTIONS:
Radiation: PET/MRI or separate PET/CT and MRI — PET/MRI or separate PET/CT and MRI using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan).
  Cohort 1 and 2 are examined twice, first one week after PCI/stent and then a second examination 2 to 8 months after the first. Cohorts 3, and 4 are examined once.

SUMMARY:
An observational, cross-sectional, longitudinal, microdosing Position Emission Tomography (PET) imaging study to investigate platelet derived growth factor receptor beta (PDGFRß) expression in the heart of patients with high or low risk of heart failure after a ST-Elevation Myocardial Infarction (STEMI) after a percutaneous coronary intervention (PCI) with a stent procedure, as well as in patients with heart failure with preserved ejection fraction (HFpEF) and healthy individuals.

DETAILED DESCRIPTION:
PDGFRß is a biomarker for pericytes which are identified as the progenitor of myofibroblast and fibroblast responsible for extra-cellular matrix proteins deposition in fibrotic heart. The Positron Emission Tomography (PET) tracer [68Ga]Ga-Dodecane tetra acetic acid (DOTA)-Cys-ATH001 is a marker for fibrogenic cells by targeting the surface receptor PDGFRß.

Four cohorts are examined by Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) or separate Positron Emission Tomography/Computed Tomography (PET/CT) and MRI using the following imaging protocol: 15O-H20 (myocardial perfusion, up to 10 min dynamic PET scan), [68Ga]Ga-DOTA-Cys-ATH001 (PDGFRß PET, up to 60 min dynamic + static full body PET scans), and Gd-MRI (extracellular volume in infarct, around 10 min MRI scan).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial and able to comply with all trial procedures and requirements.
* Male or female participant aged 40 to 70 years, inclusive, at the screening visit.
* Women of childbearing potential must practice abstinence from heterosexual intercourse or must agree to use a highly effective method of contraception.

Cohort-specific inclusion criteria:

Cohort 1, STEMI high-risk patients:

* NT-proBNP >500 pg/mL within 48 hrs after PCI
* Post-PCI Thrombolysis In Myocardial Infarction (TIMI) score <3.
* No previous history of coronary artery disease or heart failure.

Cohort 2, STEMI low-risk patients

* NT-proBNP <500 pg/mL within 48 hrs after PCI
* Post-PCI TIMI score 3.
* No previous history of coronary artery disease or heart failure.

Cohort 3 (HFpEF patients)

* Presence of signs and symptoms of HF
* Ejection Fraction ≥50%
* Elevated levels of natriuretic peptides (NT-proBNP≥125pg/mL)
* At least one of the following:
* Relevant structural heart disease (left ventricular hypertrophy or left atrial enlargement)
* Diastolic dysfunction

Cohort 4 (healthy participants)

* Individuals with no history of coronary disease or heart failure.
* Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG, and laboratory values at the time of the screening visit, as judged by the Investigator.

Exclusion Criteria:

* Any contraindication for MRI according to a standard checklist
* Having worked as a metal worker or welder.
* Contraindication for gadolinium-based contrast agents such as risk of nephrogenic systemic fibrosis (NSF) or allergy to gadolinium.
* Kidney dysfunction measured as estimated Glomerular filtration rate (eGFR)<30 mL/min/1.73m2
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial or influence the results or the participant's ability to participate in the trial.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the screening visit.
* Any malignancy within the past 12 months before the screening visit, with the exception of successfully treated basal cell carcinoma of the skin or in situ prostate cancer under active surveillance, with no interventions scheduled during the period of trial participation.
* Any active gastrointestinal hemorrhage in the past six months.
* Acute or chronic disabling stroke.
* Aortic aneurysm or aortic dissection.
* Hypertensive crisis.
* Circulatory unstable condition in need for mechanical support.
* Any planned major surgery within the duration of the trial participation.
* Participants who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
* Poor peripheral venous access, as judged by the Investigator.
* The participant has any laboratory abnormality or condition that, in the Investigator's opinion, could adversely affect the safety of the participant or impair the assessment of trial results.
* The participant is using any prohibited concomitant medications as described in the protocol, at the discretion of the Investigator.
* The Investigator considers the participant unlikely to comply with trial procedures, restrictions, and requirements.

Additional exclusion criteria for all participants (cohorts 1,2 and 4):

* History of coronary artery disease or heart failure.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients with STEMI high- and low-risk, and HFpEF will be recruited and/or identified from referral sites, by Uppsala University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PET-tracer binding in myocardium | At PET/MRI baseline, and at PET/MRI at 2-8 months after baseline (cohort 1 and 2)
  Difference in [68Ga]Ga-DOTA-Cys-ATH001 Standardized Uptake Value (SUV)mean / SUVmax / SUVtot in the whole myocardium of healthy subjects compared with STEMI high-risk and low-risk patients, and HFpEF patients.
PET-tracer binding in the infarct | At PET/MRI baseline, and at PET/MRI at 2-8 months after baseline (cohort 1 and 2)
  Difference in uptake of [68Ga]Ga-DOTA-Cys-ATH001 in the infarct, as identified by Gd-MRI compared to uptake in healthy myocardium.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Henrik Grinnemo, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No